CLINICAL TRIAL: NCT05554198
Title: Evaluating a Web Delivered Behavioral Parent Training Intervention for Rural Parents of Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021B0434; GR128585 (Other: Ohio State University)
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder; Parenting; Parenting Intervention
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The proposed study uses a single group, pre/post-test, mixed method study design with quantitative data collection at baseline and post-intervention and qualitative data collection once at post-intervention. Participants will have access to the Attend Behavior program for a full year, but intervention usage monitoring and study outcomes will be assessed until post-intervention (12-weeks post-baseline).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Intervention (Experimental): pre/post-test, mixed method study design with quantitative data collection at baseline and post-intervention and qualitative data collection once at post-intervention. Participants will have access to the Attend Behavior program for a full year, but intervention usage monitoring and study outcomes will be assessed until post-intervention (12-weeks post-baseline).
  Interventions: Behavioral: Attend Behavior Parent Training

INTERVENTIONS:
Behavioral: Attend Behavior Parent Training — Attend Behavior is a Parent Training intervention available in application form for smartphones or online. Attend Behavior consists of 12 instructional modules and it is recommended that parents complete one module a week in addition to practicing the techniques taught in that course. Each learning module typically around 30 minutes to complete and includes an introductory video to give parents an overview of the different features of the application. At the start of the intervention, parents will take an assessment that will provide information for the program to create individualized goals, plans, reinforcement agents, and even daily schedules. A HIPPA compliant clinician portal within the application allows the clinician to have real time access to monitor the parent learning progress, tracked behaviors, parental notes, and message with the parent.

SUMMARY:
For parents of children with autism spectrum disorder (ASD), the severity of the child's behavior negatively correlates with parental well-being. Parental education and support buffers stress and negative effects that some parents experience. Parents living in rural areas face several barriers to obtaining support, psychoeducation, and ASD interventions due to a lack of local resources.

This pilot study will test the acceptability, feasibility and preliminary effects of Attend Behavior, a Web-based behavioral parent training (PT) program, for parents of children with ASD in rural areas. The program goals are to decrease child problem behaviors and improve parental mental health. Methods: Parents (N = 40) of young children (2-11 years old) diagnosed with ASD will be recruited. A single group pre/post-intervention design using mixed methods will be used to determine the acceptability, feasibility, and preliminary efficacy. The effects of Attend Behavior on parent mental health will be measured. The effects of Attend Behavior on child problem behaviors will be measured. Individual interviews with the parents will take place post-intervention to ascertain perspectives on Attend Behavior. Acceptability and feasibility will also be measured using the Acceptability of Intervention, Intervention Appropriateness Measure, and the Feasibility of Intervention Measure. Effect sizes will be calculated to examine the efficacy of the intervention.

DETAILED DESCRIPTION:
There has been notable increases in the prevalence of autism spectrum disorder (ASD) both in the United States and worldwide over the past few decades. For comparison, the latest prevalence rate in the US is 1 in 54 where as just 10 years prior the rate was 1 in 110. Multiple theories have been proposed to explain the steady rise in ASD prevalence including changes in diagnostic criteria, public awareness, early screening, and etiological factors. Although there remains a significant need to improve our understanding of effective treatment for children with ASD, the science and knowledge around behavioral and psychopharmacologic interventions for the treatment of ASD has progressively grown within the past few decades. Yet, parents of children with ASD living in rural areas face additional obstacles to obtain support, resources, and services for ASD due to the lack of ASD specialists and mental health care providers in their area. Despite the similar prevalence rate of ASD between urban and rural areas, and the prevalence rate of total developmental disorders in rural areas being significantly higher, children in rural areas are less likely to see a mental health professional or receive Special Education. Parents of children with ASD also report poorer mental and physical health compared to parents of neurotypical child and parents of children with other chronic or neurodevelopmental conditions. A negative correlation has also been noted between the severity of ASD and child problem behaviors with parental mental health. Therefore, interventions aimed at decreasing the severity of child disruptive behaviors may also be beneficial to parental mental health.

Behavioral parent training (PT) programs improve child and parent outcomes for children with ASD. However, families of children with ASD face barriers in accessing PT and there is an inequity in access for families residing in rural areas. PT interventions delivered via telehealth have been examined with various treatments of children with ASD. Traditionally telehealth services have required a clinician that is highly trained in the treatment of ASD. Therefore, telehealth services may reduce geographical barriers, but it does not address the disparity of treatment providers seen throughout the US.

Attend Behavior is self-administered mobile or web-based PT intervention that educates and encourages the use of evidence-based parenting skills for children with multiple behavior problems such as hyperactivity, impulsivity, mild aggression, and emotional dysregulation. Attend Behavior includes ten modules that encompass parenting strategies to reduce disruptive child behaviors. Parents take an assessment that allows Attend Behavior to tailor the intervention material to the individual parent's needs. Attend Behavior sends automatic notifications to remind the parent to engage and apply parenting skills in their everyday life. Therefore, Attend Behavior can be used by the parent independently and other health care providers such as nurses, case managers, and primary care providers have the ability to use this intervention with parents of children with ASD without prior expertise in ASD treatment.

The purpose of the proposed study is to determine the acceptability, feasibility, and preliminary effects of the Attend Behavior PT intervention with parents residing in rural areas. To accomplish this, we will use a single-group, mixed methods pre/post-test design with rural parents (N = 40) of children (2-11 years old) with ASD. Parents will be recruited from community mental health offices and schools. Data will be collected on child problem behaviors (disruptive behaviors and child noncompliance in the home), parent mental health (parenting stress and depressive symptoms), sociodemographic variables, and intervention feasibility and acceptability. Parents will complete one module of Attend Behavior weekly for 12 weeks. Data will be collected at baseline and post-intervention (12-weeks post-baseline). Parents will complete a 1:1 interview with the study PI via phone or video conference in the post-intervention period to discuss acceptability, feasibility, and satisfaction with the intervention.

Aim 1: Evaluate the acceptability and feasibility of the Attend Behavior PT intervention with rural parents of young children with ASD. 1a. Acceptability will be assessed by the Acceptability of Intervention Measure (AIM), the Intervention Appropriateness Measure (IAM), and 1:1 interview. 2a. Feasibility will be measured with the Feasibility of Intervention Measure (FIM), intervention recruitment, retention and completion monitoring, and 1:1 interview.

Aim 2: Determine the effects of Attend Behavior on parental mental health (depression and stress) and child outcomes (disruptive behavior and noncompliance in the home) from baseline to post-intervention.

We are testing the feasibility, acceptability, and preliminary effects of the mobile and/or web-delivered PT intervention, Attend Behavior, for rural parents of children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* legal guardian of one or more children ages 2-11 years old with a formal diagnosis of ASD by parent report;
* child with ASD resides at home with the parent;
* parent age is 18 years or older;
* reside in a rural (micropolitan or noncore) county;
* access to either a smartphone with the Apple App store or Google Play store or a computer with Internet access;
* ability to read English

Exclusion Criteria:

- currently participating in another behavior Parent Training program or in the past 6-months have been enrolled in another behavior Parent Training program

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Intervention acceptability Interview | Post intervention (12 weeks post-baseline)
  1:1 semi-structured interview
Intervention feasibility | Post intervention (12 weeks post-baseline)
  Rates of completion of intervention and recruitment/retention rates
Acceptability of Intervention (AIM),Intervention Appropriateness Measure (IAM), Feasibility of Intervention (FIM) | Post intervention (12 weeks post-baseline)
  Total of 12-items answered on a Likert scale of 1 = completely disagree to 5 = completely agree, the AIM, IAM, and FIM is a brief measurement to examine implementation success

SECONDARY OUTCOMES:
Aberrant Behavior Checklist (ABC) | Baseline and Post intervention (12 weeks post-baseline)
  The ABC consists of 58 questions with five subscales: irritability, withdrawal, stereotypic behavior, hyperactivity, and inappropriate speech
Home Situations Questionnaire-Autism Spectrum Disorder (HSQ-ASD) | Baseline and Post intervention (12 weeks post-baseline)
  24-item rating where parents report yes/no if the child has been noncompliant in the past 4 weeks to a variety of situations in the home setting (e.g. "when told to brush teeth"). If the child reports the child was noncompliant in a situation within the last 4 weeks, they are prompted to rate the severity of that problem on a 1-9 Likert scale with higher scores indicating higher severity.
Patient-Reported Outcome Measurement Information System (PROMIS) Depression - Short Form 6a | Baseline and Post intervention (12 weeks post-baseline)
  6-item PROMIS short form measurement prompts participants to rate how often they have felt emotions associated with depression within the past 7 days on a scale of 1 = Never to 5 = Always
Parenting Stress Index-Short Form (PSI-SF) | Baseline and Post intervention (12 weeks post-baseline)
  36-item measurement with three domains: parental distress, parent-child dysfunctional interaction, and difficult child to yield a total stress score

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University College of Nursing, Columbus, Ohio, United States